CLINICAL TRIAL: NCT02893839
Title: Study of Sensitization to Potato in Patients Consulting at the Allergy Unit in Montpellier
Brief Title: Evaluation of Allergy to Potato in a Large Cohort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UF 9045
Record Dates: First submitted 2016-08-11; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Allergy
Keywords: Allergy; cross-reactivity; oral allergy syndrome; potato; sensitization
MeSH Terms: conditions — Hypersensitivity; Oral Allergy Syndrome

ARMS (1):
- Prick to prick (Other)
  Interventions: Other: Prick to prick test

INTERVENTIONS:
Other: Prick to prick test

SUMMARY:
Patients consulting in the Allergy Unit of the Arnaud de Villeneuve Hospital for whatever suspicion of allergy were asked to participate in the study. Besides a standard battery of respiratory allergens, native raw and cooked potato were tested by means of the prick to prick method, using a metal lancet.

ELIGIBILITY:
Inclusion criteria:

* patients aged 2 years or older
* consent obtained from patients or their parents/legal representative

Exclusion criteria:

* refusal to participate in the study
* antihistamine drugs taken before testing
* pregnant women
* vulnerable patients according to French regulation

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Rate of sensitization and allergy to potato | 35 months after the first inclusion

SECONDARY OUTCOMES:
Rate of risk factors of sensitization to raw potato | 35 months after the first inclusion
Rate of risk factors of sensitization to cooked potato | 35 months after the first inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France